CLINICAL TRIAL: NCT03084458
Title: Does Activity Feedback Increase ICD Patient Activity Levels?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ashley Burch (Other)
Collaborators: Medtronic (Industry); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor-Investigator, Ashley Burch, PI, East Carolina University
Organization: East Carolina University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR3535
Record Dates: First submitted 2017-03-09; First posted 2017-03-21 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2018-01

CONDITIONS: ICD Patients
Keywords: Increasing daily physical activity

STUDY DESIGN:
Intervention Model Description: A randomized, between subjects design will allow for comparisons between the experimental and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Once consented, recruited ICD patients will complete the baseline psychosocial and quality of life measures. At the first and final visit, a 6-minute walk test will be administered. Participants will be sent text messages to encourage physical activity. Participants will be re-assessed with psychosocial and quality of life measures at 30 and 90 days post enrollment. At the final (90 day) visit participants ICD will be interrogated to obtain accelerometer activity data.
- Fitbit (Experimental): Same as control condition. In addition, participants in the experimental group will receive a Fitbit device with full instructions and troubleshooting. These participants will be given daily step goals, which will be increased during the course of the study, and be able to monitor their progress using the Fitbit app.
  Interventions: Behavioral: Fitbit

INTERVENTIONS:
Behavioral: Fitbit — The Fitbit device will allow experimental group participant access to their daily step count.
  Arms: Fitbit

SUMMARY:
Medical device technology for use by patients is gaining popularity. Modern cardiac disease management seeks to integrate multiple device technologies and capabilities to optimize health outcomes. Fitbit, Inc. manufactures a line of wireless-enabled activity, wearable trackers that are used in conjunction with a mobile device. The Fitbit trackers use three-dimensional accelerometers to sense and record movement. This technology represents a new frontier for patients and their health care providers to understand and track physical activity in real time. The primary aim of the current project is to assess whether activity feedback using FitBit technology affects implantable cardioverter defibrillator (ICD) patient activity level as measured by the ICD accelerometer. The investigators will also examine the perceived added value of Fitbit technology to an ICD patient user experience.

Approximately 50 participants will be recruited. Participants in the experimental group (n = 25) will use the Fitbit device for 12 weeks. The experimental group will receive fitness goals (number of steps per day) to increase activity from a baseline value to a minimum of 7000 steps per day by week 9 of the intervention. Both groups will receive weekly texts messages to encourage activity. Feedback about technology satisfaction, cardiac anxiety, cardiac self-care, and health care utilization will be elicited from patients at multiple time points. Additional information will be gained about patient decision-making as participants may elect to continue Fitbit use beyond the study period; this will allow for behavioral evidence of the perceived value of adding this technology.

ELIGIBILITY:
Inclusion Criteria:

* has a Medtronic ICD
* access to a smartphone, tablet, or computer with internet access
* English speaking

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-06-11 (Actual)

PRIMARY OUTCOMES:
Does increased access to information on daily activity level (FitBit) increase device (ICD) coded total activity (step count) over usual care? | 12 weeks
  At the final study visit, the ICD will be interrogated. Accelerometer data will be captured and used as a precise measure of physical activity, specifically, steps per day.
  Analyses will be conducted to determine activity (step count) changes between groups and over time.
Does activity level feedback have a greater impact on Quality of Life (QOL) than usual care? Indices of QOL will be multiple questionnaire scores entered together in a single analysis. | 12 weeks
  Questionnaires that will be used include: Cardiac Anxiety Questionnaire, Duke Activity Status Index, Fitbit Technology Satisfaction, Florida Patient Acceptance Survey, Florida Shock Anxiety Scale, Patient Health Security, Self-Care of Heart Failure Index, and the Short-Form 12 Health Survey. Analyses will be conducted to determine quality of life changes between groups and over time from the baseline, month 1, and month 3 visits.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Burch, Principal Investigator — East Carolina Univerity; Samuel Sears, Principal Investigator — East Carolina Univerity
Locations (1):
- University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No